CLINICAL TRIAL: NCT01764009
Title: Safety and Efficacy of Intramuscular Electrotransfer of Plasmid AMEP in Patients Suffering From Advanced or Metastatic Melanoma: an Open-label Phase I/II Clinical Trial - The AIMM Study (AMEP In Metastatic Melanoma)
Brief Title: Safety and Efficacy of Intramuscular Electrotransfer of Plasmid AMEP in Patients Suffering From Advanced or Metastatic Melanoma
Acronym: AIMM
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped due to low enrolment rate.
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA2011/15/02; 2011-005538-20 (EudraCT Number)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma
Keywords: Advanced Melanoma; Metastatic Melanoma; Melanoma Stage III and IV
MeSH Terms: conditions — Melanoma | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plasmid AMEP electrotransfer in muscle (Experimental)
  Interventions: Biological: naked DNA coding for protein AMEP

INTERVENTIONS:
Biological: naked DNA coding for protein AMEP — injections 28days interval of 3 increasing doses of plasmid with electrotransfer
  Other Names: electrotransfer; electroporation

SUMMARY:
The objective of the present trial is:

* to determine the dose limiting toxicity (DLT), maximal tolerated dose (MTD) and recommended phase 2 dose (RP2D) of intramuscular electrotransferred Plasmid AMEP in patients with advanced or metastatic melanoma.
* to determine the local and general safety of intramuscular electrotransferred Plasmid AMEP
* to evaluate the efficacy of intramuscular electrotransferred Plasmid AMEP

DETAILED DESCRIPTION:
In this open-label, multicentre, dose escalation phase I study, successive cohorts of 3 patients suffering from advanced or metastatic melanoma will be electrotransferred increasing doses of Plasmid AMEP into muscle. Treatment will be repeated every 28 days until progression or limiting toxicity.

Consecutive cohorts of 3 to 6 patients will be treated with increasing doses of Plasmid AMEP at three dose levels: 0.25 mg, 1 mg and 4 mg according to an adapted 3+3 design. There will be no intra-patient dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Patient with histologically or cytologically confirmed melanoma
* Patient with unresectable advanced or metastatic (stage III or IV) melanoma
* Patient with progressive melanoma (any BRAF status is permitted) not responding or intolerant to previous treatments, including patients with asymptomatic and not rapidly progressive brain metastases.
* Patient with a minimum of one measurable lesion according to RECIST guideline 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Patient having given a written informed consent

Exclusion Criteria:

* Patient eligible for curative treatments and/or any palliative treatments with demonstrated efficacy, including current treatments for brain metastasis, and including available BRAF inhibitors as indicated for patients carrying B-RAF mutated tumours if applicable.
* Patient with history of any other cancer within five years before enrollment (except cured basal cell carcinoma or cervical cancer in situ)
* Patient with inadequate organ function, defined as:
* Platelet count < 75.103 /L (> grade 2 NCI CTCAE)
* Absolute neutrophil count < 1.109 /L (> grade 2)
* Hemoglobin < 9 g/dL
* INR increased or prolonged activated partial thromboplastin time (aPTT) upper the limit of normal (ULN) (≥ grade 1)
* Creatinine clearance < 60 mL/min (Cockcroft and Gault formula) (≥ grade 2)
* Patient with ALT > 3 ULN (≥ grade 2) or patient with symptomatic liver metastasis with ALT > 5 ULN (> grade 2)
* Serum Total Bilirubin > 1.5 ULN (≥ grade 2); Patient with Gilbert's syndrome could be included if hyperbilirubinemia ≤ 3 ULN
* Not medically controlled coagulation disorder (i.e hemophilia, protein C or S deficiency…)
* Patient with electronic pacemakers, defibrillators, or any implanted electronic device
* Any cardiac dysrhythmia (> grade 2) (i.e significant ventricular arrhythmia as persistent ventricular tachycardia and/or ventricular fibrillation; severe conduction disorders as atrio-ventricular block 2 and 3, sino-atrial block)
* Recent (less than 6 months) acute vascular diseases (i.e stroke, myocardial infarction)
* Arterial vascular disorders ≥ grade 2
* Serious, non-healed wound, ulcer or bone fracture
* Significant traumatic injury within 28 days prior to study treatment start or anticipation of the need for major surgery during study treatment
* Evidence of ongoing or active viral or bacterial infection ( i.e bacterial infection requiring IV antibiotics)
* Patient with life expectancy less than 3 months
* Prior systemic therapy or any other antineoplastic treatments within the last 4 weeks, including radiotherapy or surgery
* Patients who had participated in another clinical trial in the last 30 days prior to enrolment in the present clinical trial
* Man and woman of child-bearing age without effective contraception method during the study and for 3 months after the last administration of Plasmid AMEP (i.e oral contraception or intra-uterine device for woman; i.e condom for man)
* Pregnant or nursing women
* Any significant disease, including psychiatric and neuromuscular disease, which may affect the proper evaluation of safety or efficacy or may affect ability to give informed consent
* Patients unwilling or unable to comply with protocol requirements and scheduled visits
* For contrast enhanced ultrasound (CEUS): known contraindications to SonoVue as described in the summary product characteristics (i.e cardiac or pulmonary history, hypersensitivity to sulphur hexafluoride or to any of the components of SonoVue)
* For the part II: prophylactic phenytoin in combination with dacarbazine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety-Dose Limiting toxicity determination | 8 weeks
  Dose Limiting Toxicity (DLT) defined as any grade 4 clinical or biological event related to the study treatment and occurring during the first and second course (8 weeks) Safety parameters will be assessed according to the NCI-CTCAE v4.0 classification

SECONDARY OUTCOMES:
Safety- determination of the repeated dose | 8 weeks
  Main secondary endpoints will be safety parameters; the evaluation of efficacy parameters will allow identifying preliminary efficacy of Plasmid AMEP alone and determining the RP2D.

OTHER OUTCOMES:
tolerability | 8 weeks
  * Local tolerability of the intramuscular electrotransfer of Plasmid AMEP
  * Overall tolerability: incidence, nature and severity of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bérangère VASSEUR, M.D., Study Director — BioAlliance Pharma
Locations (4):
- France (3):
  - Gustave Roussy Institute,, Le Kremlin-Bicêtre
  - Hôpital Saint Louis. Service de dermatologie, Paris
  - CHU Nancy Hôpital Brabois, Vandœuvre-lès-Nancy
- Institute of Oncology Ljubljana, Ljubljana, Slovenia